CLINICAL TRIAL: NCT03296722
Title: Effect of a Nutritional Intervention That Incorporates the Transtheoretical Model of Motivation to Change in Healthy Eating in Patients With Cardiovascular Risk Factors: a Randomized Controlled Trial
Brief Title: Effect of a Nutritional Intervention That Incorporates the Transtheoretical Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, LILIA CASTILLO MARTINEz, Professor, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NC002
Record Dates: First submitted 2017-09-02; First posted 2017-09-28 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Adherence to Fad Diet (Symptom)

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group comprised 41 patients, which was to go once a month to receive nutritional intervention with the prescription of a hypocaloric diet on the part of the nutritionist. The control group had a monthly monitoring for 3 months.
- Intervention group (Experimental): The intervention group made up of 42 patients using the transtheoretical model and MI through sessions group and sessions individual with topics of healthy eating habits taught by a nutritionist, physical activity and exercise manual taught by a physical therapist, preparation of healthy food with menu taught by graduates in gastronomy and confrontation of barriers given by a psychologist. The intervention group had a monthly monitoring for 3 months. The diet that was prescribed to the intervention group was with the characteristics of the DASH diet.
  Interventions: Behavioral: The Transtheoretical Model

INTERVENTIONS:
Behavioral: The Transtheoretical Model — Intervention with the Transtheoretical Model, through group and individual sessions with topics of healthy eating habits taught by a dietician, physical activity and exercise manual taught by a physical therapist, preparation of healthy food with menu taught by graduates in gastronomy, confrontation of barriers given by a psychologist. This group had a monthly monitoring during 3 months. The food plan that was prescribed to the intervention group was with the characteristics of the DASH diet, according to the most recent international guides of the ACC and AHA, for the reduction of cardiovascular risk.
  Arms: Intervention group

SUMMARY:
Cardiovascular diseases are the main responsible for the global burden of disease for non-communicable diseases. Its treatment and prevention is aimed at generating changes in the habits of life; however, the percentages of non-adherence are very high. The objective of the study was to evaluate the effect of a nutritional intervention in patients with cardiovascular risk that incorporates the transtheoretical model and motivational interviews on the progression in the stages of change to improve adherence to healthy eating. Methods: the investigators included 105 patients who came to the first time at clinical nutrition service in external consultation of National Institute of Medical Sciences and Nutrition Salvador Zubirán, were randomized to intervention group or control group and the stage of change of the transtheoretical model, presence or absence of anxiety and depression, anthropometry, blood pressure, physical activity, and food frequency, to determine the quality and quantity of food intake, were evaluated. Used X² and t-test for the comparison of baseline data between groups and repeated measures ANOVA to assess differences in post-intervention.

DETAILED DESCRIPTION:
The investigators included 105 patients that were randomized to intervention group or control group. The control group comprised 41 patients, that continued with the usual intervention of Clinical Nutrition Service in external consultation, attending once a month to receive nutritional intervention with the prescription of a hypocaloric diet on the part of the nutritionist. And the intervention group made up of 42 patients using the TM and MI through sessions group and sessions individual with topics of healthy eating habits taught by a nutritionist, physical activity and exercise manual taught by a physical therapist, preparation of healthy food with menu taught by graduates in gastronomy and confrontation of barriers given by a psychologist.

Both groups had a monthly monitoring for 3 months. The diet that was prescribed to the intervention group was with the characteristics of the DASH diet, according to the most recent international guides of the ACC and AHA, for the reduction of cardiovascular risk.

Once included in the study were applied to the following questionnaires to identify the stage of change according to the TM; Hospital Anxiety and Depression Scale (HAD) to evaluate the presence of anxiety and depression; 24-hours recall of multiple steps; Food consumption frequency to determine the quantity and quality of food intake and the Rapid Assessment Physical Activity Scale (RAPA), to determine the type, duration and intensity of physical activity of the subject. In addition, we measured weight, height, waist circumference, hip, and blood pressure.

Finally were described and analyzed each of the variables according to the visits in which patients were cited.

ELIGIBILITY:
Inclusion criteria

* Men and women volunteers over the age of 18 years. Referees for first time of the various specialties and subspecialties of the INCMNSZ.
* They have e-mail, telephone or personal cell phones.
* Which could go one time every month to consultation.

Submitted at least 2 of the following comorbidities:

* Overweight or obese (BMI ≥ 25kg/m2)
* DM2 with pharmacological treatment, but without treatment with insulin.
* Hypertension (≥140/90 mmHg) with or without medication
* Waist circumference greater than 80 cm women and greater than 90 cm men
* Hypertriglyceridemia (>150 mg/dl), HDL-cholesterol <40 mg/dl in men and <50 mg/dl in women. Were selected those that have two or more cardiovascular risk factors (obesity, hypertension, DM2 or dyslipidemia.

Exclusion criteria

* Diagnosis of major depression
* Cancer
* Human immunodeficiency virus (HIV)
* Acute and chronic diseases such as renal failure (GFR ˂ 30 ml/min/1.21m2)
* Disease of liver and/or heart failure
* Respiratory disease
* Bariatric surgery
* Morbid obesity (BMI ≥40 kg/m2).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Weight | 3 months
  Weight loss

IPD SHARING:
Plan to Share IPD: No